CLINICAL TRIAL: NCT01309204
Title: Efficacy and Safety of Brinzolamide 10 mg/mL/Brimonidine 2 mg/mL Eye Drops, Suspension Compared to Brinzolamide 10 mg/mL Eye Drops, Suspension Plus Brimonidine 2 mg/mL Eye Drops, Solution in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Brinzolamide/Brimonidine Twice a Day (BID) Fixed Combination (FC) vs Brinzolamide BID Plus Brimonidine BID in Patients With Open Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-10-041; 2010-024513-31 (EudraCT Number)
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Results first posted 2014-04-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-03

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: open-angle glaucoma; ocular hypertension; OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — brinzolamide; Brimonidine Tartrate; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brinz/Brim (Experimental): Vehicle, 1 drop instilled in each eye, followed by Brinzolamide 1%/brimonidine tartrate 0.2% fixed combination ophthalmic suspension, 1 drop instilled in each eye. A 10-minute waiting period separated the instillations. Study drugs were instilled twice a day for 6 months.
  Interventions: Drug: Brinzolamide 1%/brimonidine tartrate 0.2% fixed combination ophthalmic suspension; Drug: Vehicle
- Brinz+Brim (Active Comparator): Brimonidine tartrate 0.2% ophthalmic solution, 1 drop instilled in each eye, followed by Brinzolamide 1% ophthalmic suspension, 1 drop instilled in each eye. A 10-minute waiting period separated the instillations. Study drugs were instilled twice a day for 6 months.
  Interventions: Drug: Brinzolamide 1% ophthalmic suspension; Drug: Brimonidine tartrate 0.2% ophthalmic solution

INTERVENTIONS:
Drug: Brinzolamide 1%/brimonidine tartrate 0.2% fixed combination ophthalmic suspension
  Arms: Brinz/Brim
Drug: Vehicle — Inactive ingredients used as a placebo for masking purposes
  Arms: Brinz/Brim
Drug: Brinzolamide 1% ophthalmic suspension
  Other Names: AZOPT™
  Arms: Brinz+Brim
Drug: Brimonidine tartrate 0.2% ophthalmic solution
  Arms: Brinz+Brim

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of Brinzolamide/Brimonidine fixed combination in lowering intraocular pressure (IOP) relative to each of its individual active constituents instilled concomitantly (Brinzolamide+Brimonidine) in patients with open-angle glaucoma or ocular hypertension.

DETAILED DESCRIPTION:
This study consisted of 7 visits conducted during 2 sequential phases: the screening/eligibility phase, which included a screening visit and 2 eligibility visits, and a treatment phase, which included 4 on-therapy visits conducted at Week 2, Week 6, Month 3, and Month 6 (or early exit). Following washout of any IOP-lowering medication, subjects who met all inclusion/exclusion criteria at both eligibility visits and who had IOP measurements within the specified range during this period were randomized to 1 of 2 study drug groups: Brinz/Brim or Brinz+Brim.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open-angle glaucoma or ocular hypertension and, in the opinion of the Investigator, are insufficiently controlled on monotherapy or are currently on multiple IOP-lowering medications.
* Meet qualifying IOP entry criteria.
* Able to understand and sign an informed consent form.
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Women of childbearing potential if pregnant, test positive for pregnancy at Screening visit, breastfeeding, or not in agreement to use adequate birth control methods to prevent pregnancy throughout the study.
* Severe central visual field loss.
* Can not safely undergo the initial washout period and discontinue use of all IOP-lowering ocular medication(s) for the minimum specified period prior to Eligibility Visit 1.
* Best corrected visual acuity (BCVA) score worse than 55 ETDRS letters (20/80 Snellen equivalent).
* Chronic, recurrent or severe inflammatory eye disease.
* Ocular trauma within the preceding 6 months.
* Ocular infection or inflammation within the preceding 3 months.
* Clinically significant or progressive retinal disease.
* Other ocular pathology.
* Intraocular surgery within the 6 months prior to entry.
* Ocular laser surgery within the 3 months prior to entry.
* Any abnormality preventing reliable applanation tonometry.
* Any other conditions which would make the patient, in the opinion of the Investigator, unsuitable for the study.
* Recent use of high-dose (>1 gram daily) salicylate therapy.
* Recent, current, or anticipated treatment with any medication that augments adrenergic responses, or precludes use of an alpha-adrenergic agonist.
* Other protocol-specified exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1184 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Burmaster, PhD, Study Director — Alcon Research

REFERENCES:
- [Derived] Gandolfi SA, Lim J, Sanseau AC, Parra Restrepo JC, Hamacher T. Randomized trial of brinzolamide/brimonidine versus brinzolamide plus brimonidine for open-angle glaucoma or ocular hypertension. Adv Ther. 2014 Dec;31(12):1213-27. doi: 10.1007/s12325-014-0168-y. Epub 2014 Nov 28. PMID 25430900

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 102 investigational centers in the Asia-Pacific region, Canada, Central and South America, Europe, and the United States.
Pre-assignment Details: Of the 1184 enrolled, 294 subjects did not meet inclusion/exclusion criteria and were exited from the study as screen failures prior to randomization. Of the 890 randomized, 2 subjects did not receive study medication. This reporting group includes all randomized subjects who received study medication (888), as treated.
Period: Overall Study
Arm/Group | Brinz/Brim | Brinz+Brim
Started | 452 | 436
Completed | 385 | 361
Not Completed | 67 | 75
Not completed — Adverse Event | 48 | 58
Not completed — Lost to Follow-up | 2 | 2
Not completed — Subject's decision unrelated to an AE | 9 | 10
Not completed — Inadequate control of IOP | 4 | 4
Not completed — Other | 4 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all subjects who received study medication, as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brinz/Brim | Brinz+Brim | Total
Number analyzed (Participants) | 452 | 436 | 888
Age, Customized [Number; unit: participants]
  <65 years | 227 | 211 | 438
  ≥ 65 years | 225 | 225 | 450
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 252 | 246 | 498
  Male | 200 | 190 | 390

OUTCOME MEASURES:

1. Primary Outcome: Mean Diurnal IOP Change From Baseline at Month 3
Description: Mean Diurnal IOP Change from Baseline at Month 3 (ie, the subject IOP change from baseline averaged over the 9 AM and + 2 h time points at Month 3) was measured by Goldmann applanation tonometry. The study drug was instilled approximately 15 minutes after conducting the 9AM IOP measurement. One eye from each subject was chosen as the study eye, and only data for the study eye were used for the efficacy analysis. A higher IOP can be a greater risk factor for developing glaucoma or glaucoma progression (leading to optic nerve damage).
Time Frame: Baseline (Day 1), Month 3
Population: Per Protocol (PP): All subjects who received study medication, satisfied prerandomization inclusion/exclusion criteria, and completed at least 1 scheduled on-therapy study visit. In addition, individual subject visits and data points that did not satisfy the protocol criteria may have been excluded.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | Brinz/Brim | Brinz+Brim
Number analyzed (Participants) | 384 | 373
millimeters of mercury (mmHg) | -8.5 (0.16) | -8.3 (0.16)

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were collected for the duration of the study (1 year, 8 months). An AE was defined as any untoward medical occurrence in a subject that was administered a study medication, regardless of causal relationship with the medication.
Description: This reporting group includes all subjects who received study medication, as treated. Reports of AEs were obtained through solicited and spontaneous comments from the study subjects, and through observations by the study Investigator as outlined in the study protocol.
Arm/Group | Brinz/Brim | Brinz+Brim
Serious Adverse Events (participants affected / at risk) | 11/452 | 8/436
Other Adverse Events (participants affected / at risk) | 0/452 | 0/436
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brinz/Brim (N=452) | Brinz+Brim (N=436)
Corneal erosion (Eye disorders) | 2 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0
Arthroscopy (Investigations) | 1 | 0
Finger amputation (Surgical and medical procedures) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Mastectomy (Surgical and medical procedures) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Pneumonia primary atypical (Infections and infestations) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Venous occlusion (Vascular disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.